CLINICAL TRIAL: NCT01790503
Title: An Open Label Phase 1b/2 Study of Orally Administered PLX3397 in Combination With Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Phase 1b/2 Study of PLX3397 + Radiation Therapy + Temozolomide in Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-08
Record Dates: First submitted 2013-02-07; First posted 2013-02-13 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Patients With Newly Diagnosed Glioblastoma
Keywords: glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma | interventions — pexidartinib; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1b dose escalation - 600mg/day PLX3397 cohort (Experimental): 600mg/day PLX3397, Radiation Therapy, and Temozolomide
  Interventions: Drug: PLX3397; Radiation: Radiation Therapy; Drug: Temozolomide
- Phase 1b dose escalation - 800mg/day PLX3397 (Experimental): 800mg/day PLX3397, Radiation Therapy, and Temozolomide
  Interventions: Drug: PLX3397; Radiation: Radiation Therapy; Drug: Temozolomide
- Phase 1b dose escalation - 1000 mg/day PLX3397 cohort (Experimental): 1000 mg/day PLX3397, Radiation Therapy, and Temozolomide
  Interventions: Drug: PLX3397; Radiation: Radiation Therapy; Drug: Temozolomide
- Phase 2 - Recommended phase 2 dose of PLX3397 (Experimental): Recommended phase 2 dose of PLX3397 (800mg/day), Radiation therapy, and Temozolomide
  Interventions: Drug: PLX3397; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Drug: PLX3397
  Other Names: Pexidartinib
Radiation: Radiation Therapy
Drug: Temozolomide
  Other Names: TMZ; Temodar

SUMMARY:
The study objectives are to assess the potential for PLX3397 to improve the efficacy of standard of care radiation therapy (RT) + temozolomide in patients with newly diagnosed glioblastoma (GBM).

DETAILED DESCRIPTION:
Study drug will be administered twice daily for 7 days prior to the initiation of RT (radiation therapy)and will continue twice daily during the course of RT. The RT schedule will be once daily for 5 days per week for 6 weeks (total radiation dose of 60 Gy. Oral temozolomide will be administered once daily (7 days per week) for the duration of RT. Four weeks after the completion of the course of RT, patients will be started on once-daily adjuvant temozolomide (Day 1-5 of a 28 day cycle) and PLX3397 twice daily (28 days of a 28 day cycle) for up to 12 cycles in the absence of progressive disease or unacceptable toxicities. After discontinuation of study drug, patients will continue to be followed for OS every 6 months. For patients participating in the run-in Phase 1b of the study, intra patient dose escalation will be permitted after a RP2D has been established. The Phase 2 portion of the study will enroll patients to be treated with PLX3397 at RP2D.

For the Phase 1b portion of the study, 2 cohorts (800 mg/day and 1000 mg/day) are planned to be enrolled at approximately 7-10 sites. Each cohort will consist of approximately 7 patients. Therefore, a minimum of 14 patients are planned to be enrolled in Phase 1b. Additional patients may be required for replacement patients, or if lower dose cohorts (600 mg or 400 mg) are required. For the Phase 2 portion of the study, enrollment is planned to include approximately 44 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years old.
* Histologically confirmed definitive GBM or gliosarcoma by partial or complete surgical resection (i.e. not by biopsy only) within 5 weeks prior to PLX3397 administration (C1D1). Tumor must have a supratentorial component. For all patients, availability of a surgical paraffin tumor block sufficient to generate at least 20 unstained slides; or, if a paraffin tumor block is unavailable, at least 20 unstained slides.
* The patient must have recovered from the effects of surgery, post-operative infection, and other complications before study registration.
* A diagnostic contrast-enhanced MRI or CT scan of the brain must be performed preoperatively and postoperatively prior to the initiation of radiotherapy, within 28 days (preferably 14 days) prior to C1D1.
* Patients unable to undergo MR imaging because of non-compatible devices can be enrolled, provided pre- and post-operative contrast-enhanced CT scans are obtained and are of sufficient quality.
* Patients must receive RT at the participating institution.
* Women of child-bearing potential must have a negative pregnancy test within 14 days of initiation of dosing and must agree to use an acceptable method of birth control while on study drug and for 3 months after the last dose. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year. Men of child-bearing potential must also agree to use an acceptable method of birth control while on study drug, and for 3 months after the last dose.
* Karnofsky performance status of ≥70.
* Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥1.5x 109/L, Hgb >10 g/dL, platelet count ≥100 x 109/L, AST/ALT ≤2.5x ULN, creatinine ≤1.5x ULN).
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.

Exclusion Criteria:

* Evidence of recurrent GBM or metastases detected outside of the cranial vault.
* Investigational drug use within 28 days of the first dose of PLX3397 or concurrently.
* Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment.
* Prior radiation or chemotherapy for glioblastoma or glioma.
* Prior chemotherapy or radiosensitizers for cancer of the head and neck (except for T1 glottic cancer) that would result in an overlap of radiation fields.
* Prior allergic reaction to temozolomide.
* History of Grade 2 (CTCAE v4) or greater acute intracranial hemorrhage.
* Active cancer (either concurrent or within the last 3 years) that requires non-surgical therapy (e.g. chemotherapy or radiation therapy), with the exception of surgically treated basal or squamous cell carcinoma of the skin, melanoma in-situ, or carcinoma in-situ of the cervix.
* Chronic active hepatitis B or C.
* Refractory nausea and vomiting, malabsorption, biliary shunt, or significant bowel resection that would preclude adequate absorption of study drug.
* Patients with serious illnesses, uncontrolled infection, medical conditions, or other medical history including abnormal laboratory results, which in the investigator's opinion would be likely to interfere with a patient's participation in the study, or with the interpretation of the results.
* Women of child-bearing potential who are pregnant or breast feeding.
* At Screening QTcF ≥450 msec for males and ≥470 msec for females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (9):
- United States (9):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - James Cancer Hospital/Ohio State University, Columbia, Ohio
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Result] Gilbert MR, Wang M, Aldape KD, Stupp R, Hegi ME, Jaeckle KA, Armstrong TS, Wefel JS, Won M, Blumenthal DT, Mahajan A, Schultz CJ, Erridge S, Baumert B, Hopkins KI, Tzuk-Shina T, Brown PD, Chakravarti A, Curran WJ Jr, Mehta MP. Dose-dense temozolomide for newly diagnosed glioblastoma: a randomized phase III clinical trial. J Clin Oncol. 2013 Nov 10;31(32):4085-91. doi: 10.1200/JCO.2013.49.6968. Epub 2013 Oct 7. PMID 24101040
- [Result] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 participants (22 in Phase 1b; 43 in Phase 2) who met all inclusion criteria and no exclusion criteria were enrolled and treated in the study at 10 clinic sites in the United States.
Pre-assignment Details: This study included Phase 1b dose escalation where 5 cohorts were planned to be enrolled, each with approximately 7 participants (3+3 design) and Phase 2 where 37 participants were planned to be enrolled with the 7 participants treated at the RP2D level determined in the Phase 1b dose escalation phase yielding approximately 44 participants.
Groups:
- Phase 1b Dose Escalation - 600 mg/600 mg: Participants received 600 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks), followed by 600 mg/day PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 600 mg/800 mg: Participants received 600 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks), followed by 800 mg/day PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter
- Phase 1b Dose Escalation - 600 mg/1000 mg: Participants received 600 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks), followed by 1000 mg/day PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 600 mg: Participants received 600 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks). No adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 800 mg/1000 mg: Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (5 days per week for six weeks) followed by 1000 mg PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 800 mg (5 Days); Phase 2 - 800 mg: Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (5 days per week for six weeks). No adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 800 mg/600 mg: Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks) followed by 600 mg/day PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 800 mg/800 mg: Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks) followed by 800 mg/day PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter.
- Phase 1b Dose Escalation - 800 mg (7 Days): Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks) No adjuvant therapy thereafter.
- Phase 2 - 800 mg/800 mg: Participants received 800 mg/day PLX3397 in combination with radiation therapy, and temozolomide (5 days per week for six weeks) followed by 800 mg/day PLX3397 (daily dosing) and temozolomide (once daily on days 1-5 of each 28 day cycle) adjuvant therapy thereafter.
Period: Overall Study
Arm/Group | Phase 1b Dose Escalation - 600 mg/600 mg | Phase 1b Dose Escalation - 600 mg/800 mg | Phase 1b Dose Escalation - 600 mg/1000 mg | Phase 1b Dose Escalation - 600 mg | Phase 1b Dose Escalation - 800 mg/1000 mg | Phase 1b Dose Escalation - 800 mg (5 Days) | Phase 1b Dose Escalation - 800 mg/600 mg | Phase 1b Dose Escalation - 800 mg/800 mg | Phase 1b Dose Escalation - 800 mg (7 Days) | Phase 2 - 800 mg/800 mg | Phase 2 - 800 mg
Started | 3 | 1 | 1 | 2 | 5 | 5 | 1 | 1 | 3 | 27 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 3 | 1 | 1 | 2 | 5 | 5 | 1 | 1 | 3 | 26 | 16
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 4 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Disease progression | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 17 | 7
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Non Compliance | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b Dose Escation - 800 mg (7 Days): Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks) No adjuvant therapy thereafter.
- Total: Total of all reporting groups
Arm/Group | Phase 1b Dose Escalation - 600 mg/600 mg | Phase 1b Dose Escalation - 600 mg/800 mg | Phase 1b Dose Escalation - 600 mg/1000 mg | Phase 1b Dose Escalation - 600 mg | Phase 1b Dose Escalation - 800 mg/1000 mg | Phase 1b Dose Escalation - 800 mg (5 Days) | Phase 1b Dose Escalation - 800 mg/600 mg | Phase 1b Dose Escalation - 800 mg/800 mg | Phase 1b Dose Escation - 800 mg (7 Days) | Phase 2 - 800 mg/800 mg | Phase 2 - 800 mg | Total
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 5 | 5 | 1 | 1 | 3 | 27 | 16 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 0 | 2 | 5 | 4 | 0 | 1 | 3 | 7 | 11 | 37
  >=65 years | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 20 | 5 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (6.4) | 23.0 (0) | 73 (0) | 48.0 (17.0) | 50.8 (15.7) | 60.8 (8.6) | 30.0 (0) | 51.0 (0) | 53.3 (4.2) | 55.7 (10.8) | 59.0 (10.7) | 55.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 8 | 7 | 24
  Male | 1 | 1 | 1 | 1 | 3 | 2 | 0 | 1 | 3 | 19 | 9 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 0 | 2 | 3 | 4 | 1 | 1 | 3 | 25 | 16 | 58
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 1 | 2 | 5 | 5 | 1 | 1 | 3 | 27 | 16 | 65

OUTCOME MEASURES:

1. Primary Outcome: Summary of the Median Progression-free Survival (mPFS) in the Combined 800 mg, 5 Days/Week Dose Group
Description: Progression was determined by Response Assessment in Neuro-Oncology (RANO) criteria and progression-free survival (PFS) was analyzed based on the non-parametric Kaplan-Meier method.
Time Frame: Assessed from date of first dose administered to date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years 4 months.
Population: mPFS was assessed in the modified intent-to-treat RP2D and the per protocol (PP) populations.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Combined 800 mg, 5 Days/Week: All participants in Phase 1b or 2 who received 800 mg/day PLX3397 (5 days/week) during combination therapy.
Arm/Group | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 53
months
  mITT RP2D: number analyzed (Participants) | 52
  mITT RP2D | 6.7 [4.5 to 11.5]
  PP RP2D: number analyzed (Participants) | 38
  PP RP2D | 6.9 [4.5 to 10.3]

2. Primary Outcome: Summary of the Median Progression-free Survival (mPFS) in the Study Group Compared With Historical Control From Medical Literature
Description: mPFS was based on model parameters estimated by maximum likelihood with a Newton-Raphson algorithm. The Radiation Therapy Oncology Group (RTOG) 0525 study was the main historical control used for statistical analysis. Additionally, RTOG-0825 was also used to support this outcome measure.
Time Frame: as for outcome 1
Population: mPFS was based on model parameters estimated by maximum likelihood with a Newton-Raphson algorithm. The Radiation Therapy Oncology Group (RTOG) 0525 study was the main historical control.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- RP2D: mPFS was assessed in the RP2D population at Cycle 1, Day 1.
- RP2D-0525 (Cycle 1, Day 1): mPFS was assessed in the RP2D population in the RTOG 0525 study at Cycle 1, Day 1.
- RP2D-0825: mPFS was assessed in the RP2D population in the RTOG 0825 study at Cycle 2, Day 1.
- RP2D-0525 (Rest Period, Day 15): mPFS was assessed in the RP2D population in the RTOG 0525 study at the Rest Period, Day 15.
Arm/Group | RP2D | RP2D-0525 (Cycle 1, Day 1) | RP2D-0825 | RP2D-0525 (Rest Period, Day 15)
Number analyzed (Participants) | 53 | 43 | 49 | 43
months | 7.7 [5.6 to 10.4] | 7.6 [5.5 to 10.6] | 7.0 [5.1 to 9.5] | 6.1 [4.4 to 8.5]
Statistical Analysis 1: Comparison: RP2D vs RP2D-0525 (Cycle 1, Day 1); Test type: Other; p = 0.456, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.71 to 1.36]
Statistical Analysis 2: Comparison: RP2D vs RP2D-0825; Test type: Other; p = 0.619, Log Rank; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.77 to 1.43]
Statistical Analysis 3: Comparison: RP2D vs RP2D-0525 (Rest Period, Day 15); Test type: Other; p = 0.272, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.65 to 1.26]

3. Secondary Outcome: Summary of the Median Progression-free Survival (mPFS) by Subgroups in the Modified Intent-To-Treat Population on the Recommended Phase 2 Dose
Description: Progression was determined by Response Assessment in Neuro-Oncology (RANO) criteria and progression-free survival (PFS) was analyzed based on the non-parametric Kaplan-Meier method. mPFS was analyzed by age group, extent of surgery, baseline Karnofsky Performance Status (KPS), and O6-methylguanine-DNA methyltransferase status (MGMT).
  The scale range for the baseline Karnofsky Performance Status is from 0-100, with 0 indicating that the participant is dead and 100 indicating that the participant is Normal no complaints, no evidence of disease. The higher the number, the better the outcome.
Time Frame: as for outcome 1
Population: mPFS was assessed in the mITT RP2D population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 53
months
  Age: 18-64 years: number analyzed (Participants) | 39
  Age: 18-64 years | 6 [4.5 to 12.4]
  Age: 65+ years: number analyzed (Participants) | 13
  Age: 65+ years | 10 [2.7 to 11.5]
  Extent of surgery: complete resection: number analyzed (Participants) | 23
  Extent of surgery: complete resection | 6 [4.2 to 12.3]
  Extent of surgery: partial resection: number analyzed (Participants) | 26
  Extent of surgery: partial resection | 9 [4.5 to 15.4]
  Baseline KPS: 70-89: number analyzed (Participants) | 18
  Baseline KPS: 70-89 | 4 [2.6 to 4.5]
  Baseline KPS: 90-100: number analyzed (Participants) | 34
  Baseline KPS: 90-100 | 11 [6.2 to 14.7]
  MGMT status: methylated: number analyzed (Participants) | 23
  MGMT status: methylated | 10 [5.2 to 15.4]
  MGMT status: unmethylated: number analyzed (Participants) | 27
  MGMT status: unmethylated | 4 [3.9 to 10.2]
Statistical Analysis 1: Comparison: Combined 800 mg, 5 Days/Week; Comparison between age subgroups: 18-64 years vs 65+ years; Test type: Other; p = 0.440, t-test, 2 sided
Statistical Analysis 2: Comparison: Combined 800 mg, 5 Days/Week; Comparison between extent of surgery subgroups: complete resection vs partial resection; Test type: Other; p = 0.699, t-test, 2 sided
Statistical Analysis 3: Comparison: Combined 800 mg, 5 Days/Week; Comparison between baseline KPS subgroups: 70-89 vs 90-100; Test type: Other; p = 0.003, t-test, 2 sided
Statistical Analysis 4: Comparison: Combined 800 mg, 5 Days/Week; Comparison between MGMT status subgroups: methylated vs unmethylated; Test type: Other; p = 0.201, t-test, 2 sided

4. Secondary Outcome: Summary of the Overall Survival in The Study Population
Description: Overall Survival (OS) was defined as the number of days from the first day of treatment (C1D1) to the date of death and analyzed using a non-parametric Kaplan Meier method.
Time Frame: Assessed from date of first dose administered to date of death from any cause, assessed up to 4 years 4 months
Population: OS was assessed in the mITT RP2D and PP RP2D populations.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 53
months
  mITT RP2D | 13.1 [11.5 to 24.5]
  PP RP2D: number analyzed (Participants) | 38
  PP RP2D | 12.4 [9.9 to NA] — In Kaplan-Meier analysis, the upper limit of median survival's confidence interval is non-estimable (NE) when the upper confidence interval curve does not drop to or below the 50% line

5. Secondary Outcome: Summary of the Overall Survival in the Study Group Compared With Historical Control From Medical Literature
Description: Overall Survival was calculated using a parametric model. The Radiation Therapy Oncology Group (RTOG) 0525 study was the main historical control used for statistical analysis. Additionally, RTOG-0825 was also used to support this outcome measure
Time Frame: Assessed from date of first dose administered to the date of death from any cause, assessed up to 4 years 4 months.
Population: Median OS was based on model parameters estimated by maximum likelihood with a Newton-Raphson algorithm. The Radiation Therapy Oncology Group (RTOG) 0525 study was the main historical control.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- RP2D: OS was assessed in the RP2D population at Cycle 1, Day 1.
- RP2D-0525 (Cycle 1, Day 1): OS was assessed in the RP2D population in the RTOG 0525 study at Cycle 1, Day 1.
- RP2D-0825: OS was assessed in the RP2D population in the RTOG 0825 study at Cycle 2, Day 1.
- RP2D-0525 (Rest Period, Day 15): OS was assessed in the RP2D population in the RTOG 0525 study at the Rest Period, Day 15.
Arm/Group | RP2D | RP2D-0525 (Cycle 1, Day 1) | RP2D-0825 | RP2D-0525 (Rest Period, Day 15)
Number analyzed (Participants) | 53 | 43 | 49 | 43
months | 18.8 [12.6 to 28.0] | 20.2 [12.9 to 31.6] | 17.0 [11.3 to 25.6] | 16.9 [10.8 to 26.5]
Statistical Analysis 1: Comparison: RP2D vs RP2D-0525 (Cycle 1, Day 1); Test type: Other; p = 0.389, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.60 to 1.47]
Statistical Analysis 2: Comparison: RP2D vs RP2D-0825; Test type: Other; p = 0.393, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.63 to 1.42]
Statistical Analysis 3: Comparison: RP2D vs RP2D-0525 (Rest Period, Day 15); Test type: Other; p = 0.469, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.63 to 1.54]

6. Secondary Outcome: Summary of the Overall Survival by Subgroups in the Modified Intent-To-Treat Population on the Recommended Phase 2 Dose
Description: Overall Survival was calculated using a non-parametric Kaplan-Meier analysis method. Median OS was analyzed by age group, extent of surgery, baseline Karnofsky Performance Status (KPS), and O6-methylguanine-DNA methyltransferase status (MGMT).
  The scale range for the baseline Karnofsky Performance Status is from 0-100, with 0 indicating that the participant is dead and 100 indicating that the participant is Normal no complaints, no evidence of disease. The higher the number, the better the outcome.
Time Frame: Assessed from date of first dose administered to the date of death from any cause, assessed up to 4 years 4 months.
Population: OS was assessed in the mITT RP2D population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 53
months
  Age group: 18-64 years: number analyzed (Participants) | 40
  Age group: 18-64 years | 14.3 [12.3 to NA] — In Kaplan-Meier analysis, the upper limit of median survival's confidence interval is non-estimable (NE) when the upper confidence interval curve does not drop to or below the 50% line
  Age group: 65+ years: number analyzed (Participants) | 13
  Age group: 65+ years | 11 [4.3 to 24.5]
  Extent of surgery: complete resection: number analyzed (Participants) | 23
  Extent of surgery: complete resection | 14 [9.9 to 24.5]
  Extent of surgery: partial resection: number analyzed (Participants) | 27
  Extent of surgery: partial resection | 13 [7.9 to 13]
  Basline KPS: 70-89: number analyzed (Participants) | 18
  Basline KPS: 70-89 | 8 [6.9 to 12.4]
  Baseline KPS: 90-100: number analyzed (Participants) | 35
  Baseline KPS: 90-100 | 24 [13.1 to 24]
  MGMT status: methylated: number analyzed (Participants) | 23
  MGMT status: methylated | 15 [9.7 to 15]
  MGMT: unmethylated: number analyzed (Participants) | 27
  MGMT: unmethylated | 12 [7.9 to 20.7]
Statistical Analysis 1: Comparison: Combined 800 mg, 5 Days/Week; Comparison between age subgroups: 18-64 years vs 65+ years; Test type: Other; p = 0.063, t-test, 2 sided
Statistical Analysis 2: Comparison: Combined 800 mg, 5 Days/Week; Comparison between extent of surgery subgroups: complete resection vs partial resection; Test type: Other; p = 0.969, t-test, 2 sided
Statistical Analysis 3: Comparison: Combined 800 mg, 5 Days/Week; Comparison between baseline KPS subgroups: 70-89 vs 90-100; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Combined 800 mg, 5 Days/Week; Comparison between MGMT status subgroups: methylated vs unmethylated; Test type: Other; p = 0.501, t-test, 2 sided

7. Secondary Outcome: Summary of Best Overall Response by Subgroups in the Modified Intent-To-Treat Population on the Recommended Phase 2 Dose
Description: Best Overall Response (based on the RANO response) was defined as the highest overall response recorded from the start of study treatment until the end of treatment. Per the Response Assessment in Neuro-Oncology (RANO) criteria for measurable lesions and assessed by Cranial MRI scan, summarized as: Complete Response (CR), Disappearance of all enhancing disease (measurable and non-measurable); Partial Response (PR), >=50% decrease of all measurable enhancing lesions; Stable disease, does not qualify for complete response, partial response, or progression, and progression, >25% increase in enhancing lesions despite stable or increasing steroid use or any new lesions.
Time Frame: Assessed from Baseline and every 8 weeks, up to 4 years 4 months
Population: Best Overall Response was assessed in the mITT RP2D population.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 53
Participants
  Age group: 18-64 years: number analyzed (Participants) | 39
  Age group: 18-64 years: Complete response (CR) | 2
  Age group: 18-64 years: Partial response (PR) | 4
  Age group: 18-64 years: CR+PR | 6
  Age group: 18-64 years: Stable disease | 18
  Age group: 18-64 years: Progressive disease | 9
  Age group: 18-64 years: Unable to access | 0
  Age group: 18-64 years: Unknown | 0
  Age group: 65+ years: number analyzed (Participants) | 11
  Age group: 65+ years: Complete response (CR) | 0
  Age group: 65+ years: Partial response (PR) | 1
  Age group: 65+ years: CR+PR | 1
  Age group: 65+ years: Stable disease | 6
  Age group: 65+ years: Progressive disease | 3
  Age group: 65+ years: Unable to access | 0
  Age group: 65+ years: Unknown | 0
  Complete resection: number analyzed (Participants) | 21
  Complete resection: Complete response (CR) | 1
  Complete resection: Partial response (PR) | 2
  Complete resection: CR+PR | 3
  Complete resection: Stable disease | 10
  Complete resection: Progressive disease | 5
  Complete resection: Unable to access | 0
  Complete resection: Unknown | 0
  Partial resection: number analyzed (Participants) | 27
  Partial resection: Complete response (CR) | 1
  Partial resection: Partial response (PR) | 3
  Partial resection: CR+PR | 4
  Partial resection: Stable disease | 13
  Partial resection: Progressive disease | 6
  Partial resection: Unable to access | 0
  Partial resection: Unknown | 0
  Baseline KPS: 70-89: number analyzed (Participants) | 17
  Baseline KPS: 70-89: Complete response (CR) | 0
  Baseline KPS: 70-89: Partial response (PR) | 1
  Baseline KPS: 70-89: CR+PR | 1
  Baseline KPS: 70-89: Stable disease | 7
  Baseline KPS: 70-89: Progressive disease | 8
  Baseline KPS: 70-89: Unable to access | 0
  Baseline KPS: 70-89: Unknown | 0
  Baseline KPS: 90-100: number analyzed (Participants) | 33
  Baseline KPS: 90-100: Complete response (CR) | 2
  Baseline KPS: 90-100: Partial response (PR) | 4
  Baseline KPS: 90-100: CR+PR | 6
  Baseline KPS: 90-100: Stable disease | 17
  Baseline KPS: 90-100: Progressive disease | 4
  Baseline KPS: 90-100: Unable to access | 0
  Baseline KPS: 90-100: Unknown | 0
  MGMT status: methylated: number analyzed (Participants) | 22
  MGMT status: methylated: Complete response (CR) | 1
  MGMT status: methylated: Partial response (PR) | 3
  MGMT status: methylated: CR+PR | 4
  MGMT status: methylated: Stable disease | 11
  MGMT status: methylated: Progressive disease | 3
  MGMT status: methylated: Unable to access | 0
  MGMT status: methylated: Unknown | 0
  MGMT status: unmethylated: number analyzed (Participants) | 27
  MGMT status: unmethylated: Complete response (CR) | 1
  MGMT status: unmethylated: Partial response (PR) | 2
  MGMT status: unmethylated: CR+PR | 3
  MGMT status: unmethylated: Stable disease | 12
  MGMT status: unmethylated: Progressive disease | 9
  MGMT status: unmethylated: Unable to access | 0
  MGMT status: unmethylated: Unknown | 0
Statistical Analysis 1: Comparison: Combined 800 mg, 5 Days/Week; Comparison between age subgroups: 18-64 years vs 65+ years; Test type: Other; p = 0.705, t-test, 2 sided
Statistical Analysis 2: Comparison: Combined 800 mg, 5 Days/Week; Comparison between extent of surgery subgroups: complete resection vs partial resection; Test type: Other; p > 0.999, t-test, 2 sided
Statistical Analysis 3: Comparison: Combined 800 mg, 5 Days/Week; Comparison between baseline KPS subgroups: 70-89 vs 90-100; Test type: Other; p = 0.099, t-test, 2 sided
Statistical Analysis 4: Comparison: Combined 800 mg, 5 Days/Week; Comparison between MGMT status subgroups: methylated vs unmethylated; Test type: Other; p = 0.348, t-test, 2 sided

8. Secondary Outcome: Overview of Most Frequent System Organ Classes Reported in Phase 1b of the Modified Intent-To-Treat Population
Time Frame: Baseline up to 30 days after last dose, up to 4 years 4 months
Population: Safety was assessed in the mITT population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Dose Escalation - 800 mg; Phase 1b Dose Escation - 800 mg: Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (5 days per week for six weeks). No adjuvant therapy thereafter.
Arm/Group | Phase 1b Dose Escalation - 600 mg/600 mg | Phase 1b Dose Escalation - 600 mg/800 mg | Phase 1b Dose Escalation - 600 mg/1000 mg | Phase 1b Dose Escalation - 600 mg | Phase 1b Dose Escalation - 800 mg/1000 mg | Phase 1b Dose Escalation - 800 mg | Phase 1b Dose Escalation - 800 mg/600 mg | Phase 1b Dose Escalation - 800 mg/800 mg | Phase 1b Dose Escation - 800 mg
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 5 | 5 | 1 | 1 | 3
Participants
  General Disorders and Administrative Site | 2 | 0 | 1 | 1 | 5 | 5 | 1 | 1 | 3
  Nervous System Disorders | 3 | 1 | 1 | 2 | 5 | 4 | 1 | 0 | 2
  Skin and Subcutaneous Tissue Disorders | 3 | 1 | 1 | 2 | 5 | 4 | 0 | 1 | 1
  Gastrointestinal Disorders | 3 | 1 | 1 | 1 | 5 | 3 | 0 | 0 | 2
  Metabolism and Nutrition Disorders | 3 | 1 | 1 | 1 | 4 | 2 | 0 | 1 | 2
  Psychiatric Disorders | 2 | 1 | 1 | 2 | 3 | 1 | 1 | 0 | 1
  Infections and Infestations | 1 | 0 | 1 | 1 | 5 | 1 | 0 | 0 | 3
  Investigations | 1 | 0 | 1 | 1 | 4 | 2 | 1 | 0 | 3
  Respiratory, Thoracic, and Mediastinal Disorders | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 2
  Musculoskeletal and Connective Tissue Disorders | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 1
  Blood and Lymphatic Tissue Disorders | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1
  Vascular Disorders | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 2
  Renal and Urinary Disorders | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1
  Eye Disorders | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
  Injury, Poisoning, and Procedural Complications | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Ear and Labyrinth | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Endocrine Disorders | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Cardiac Disorders | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hepatobiliary Disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Reproductive System and Breast Disorders | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Immune System Disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neoplasms Benign, Malignant, and Unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Overview of Most Frequent System Organ Classes Reported in Phase 2 of the Modified Intent-To-Treat Population
Time Frame: Baseline up to 30 days after last dose, up to 4 years 4 months
Population: Safety was assessed in the mITT population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Total: All participants in Phase 2 who received 800 mg/day PLX3397 in combination therapy.
Arm/Group | Phase 2 - 800 mg/800 mg | Phase 2 - 800 mg | Phase 2 Total | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 27 | 16 | 43 | 53
Participants
  General Disorders and Administration Site | 24 | 13 | 37 | 47
  Skin and Subcutaneous Tissue Disorders | 24 | 12 | 36 | 45
  Nervous System Disorders | 22 | 12 | 34 | 43
  Gastrointestinal Disorders | 21 | 12 | 33 | 41
  Metabolism and Nutrition Disorders | 16 | 8 | 24 | 30
  Psychiatric Disorders | 17 | 6 | 23 | 27
  Investigations | 12 | 9 | 21 | 27
  Musculoskeletal and Connective Tissue Disorders | 13 | 7 | 20 | 25
  Blood and Lymphatic System Disorders | 14 | 2 | 16 | 18
  Injury, Poisoning, and Procedural Complications | 10 | 6 | 16 | 18
  Eye Disorders | 7 | 6 | 13 | 16
  Vascular Disorders | 9 | 4 | 13 | 18
  Respiratory, Thoracic, and Mediastinal Disorders | 7 | 3 | 10 | 16
  Renal and Urinary Disorders | 7 | 2 | 9 | 13
  Cardiac Disorders | 5 | 2 | 7 | 8
  Endocrine Disorders | 5 | 1 | 6 | 7
  Ear and Labyrinth Disorders | 3 | 1 | 4 | 5
  Reproductive System and Breast Disorders | 2 | 0 | 2 | 3
  Neoplasms Benign, Malignant, and Unspecified | 2 | 0 | 2 | 2
  Hepatobiliary Disorders | 0 | 1 | 1 | 1
  Immune System Disorders | 1 | 0 | 1 | 1

10. Secondary Outcome: Number of Patients With Clinically Significant Abnormal Chemistry and Hematology Values Reported as Adverse Events by Preferred Term in Phase 1b of the Modified Intent-To-Treat Population
Time Frame: Baseline up to 30 days after last dose, up to 4 years 4 months
Population: Abnormal chemistry and hematology values were assessed in the mITT population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Dose Escation - 800 mg (No Adjuvant Therapy): Participants received 800 mg/day PLX3397 in combination with radiation therapy and temozolomide (7 days per week for six weeks) No adjuvant therapy thereafter.
Arm/Group | Phase 1b Dose Escalation - 600 mg/600 mg | Phase 1b Dose Escalation - 600 mg/800 mg | Phase 1b Dose Escalation - 600 mg/1000 mg | Phase 1b Dose Escalation - 600 mg | Phase 1b Dose Escalation - 800 mg/1000 mg | Phase 1b Dose Escalation - 800 mg (5 Days) | Phase 1b Dose Escalation - 800 mg/600 mg | Phase 1b Dose Escalation - 800 mg/800 mg | Phase 1b Dose Escation - 800 mg (No Adjuvant Therapy)
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 5 | 5 | 1 | 1 | 3
Participants
  Thrombocytopenia | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
  Neutropenia | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Anaemia | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Lymphopenia | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AST increased | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Neutrophil count decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Leukopenia | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Febrile neutropenia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  ALT increased | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Bone marrow failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Haemolysis | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

11. Secondary Outcome: Number of Patients With Clinically Significant Abnormal Chemistry and Hematology Values Reported as Adverse Events by Preferred Term in Phase 2, the Combined RP2D Groups in Phase 1b, and in the Study Overall Modified Intent-To-Treat Population
Time Frame: Baseline up to 30 days after last dose, up to 4 years 4 months
Population: Abnormal chemistry and hematology values were assessed in the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - 800 mg/800 mg | Phase 2 - 800 mg | Phase 2 Total | Combined 800 mg, 5 Days/Week
Number analyzed (Participants) | 27 | 16 | 43 | 53
Participants
  Neutropenia | 6 | 1 | 7 | 9
  Thrombocytopenia | 3 | 1 | 4 | 6
  Anaemia | 5 | 1 | 6 | 7
  ALT increased | 2 | 5 | 7 | 8
  AST increased | 2 | 4 | 6 | 8
  Platelet count decreased | 4 | 1 | 5 | 7
  Lymphopenia | 2 | 1 | 3 | 4
  White blood cell count decreased | 4 | 1 | 5 | 5
  Neutrophil count decreased | 2 | 0 | 2 | 2
  Leukopenia | 1 | 1 | 2 | 2
  Febrile neutropenia | 0 | 1 | 1 | 2
  Lymphocyte count decreased | 1 | 1 | 2 | 3
  Blood alkaline phosphatase increased | 0 | 3 | 3 | 3
  Blood creatinine increased | 2 | 1 | 3 | 3
  DRESS | 0 | 1 | 1 | 1
  Liver function test abnormal | 0 | 1 | 1 | 1
  Bone marrow failure | 0 | 0 | 0 | 0
  Haemolysis | 0 | 0 | 0 | 1
  Blood bilirubin increased | 0 | 1 | 1 | 1
  Blood iron decreased | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 30 days after the last dose, up to 4 years 4 months.
Description: Adverse events that emerge (or worsen) after the first dose of study drug and within 28 days after the last dose.
  For the Other (Not Including Serious) Adverse Events data reported, data available are AEs who meet the Common Toxicity Criteria for Adverse Events (CTCAE) >=3 criteria (which is for severity, rather than frequency).
Arm/Group | Phase 1b Dose Escalation - 600 mg/600 mg | Phase 1b Dose Escalation - 600 mg/800 mg | Phase 1b Dose Escalation - 600 mg/1000 mg | Phase 1b Dose Escalation - 600 mg | Phase 1b Dose Escalation - 800 mg/1000 mg | Phase 1b Dose Escalation - 800 mg (5 Days) | Phase 1b Dose Escalation - 800 mg/600 mg | Phase 1b Dose Escalation - 800 mg/800 mg | Phase 1b Dose Escation - 800 mg (7 Days) | Phase 2 - 800 mg/800 mg | Phase 2 - 800 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/1 | 0/2 | 0/5 | 0/5 | 0/1 | 0/1 | 0/3 | 1/27 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1 | 0/1 | 2/2 | 2/5 | 2/5 | 0/1 | 0/1 | 3/3 | 13/27 | 9/16
Other Adverse Events (participants affected / at risk) | 1/3 | 1/1 | 1/1 | 2/2 | 5/5 | 5/5 | 0/1 | 1/1 | 3/3 | 18/27 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose Escalation - 600 mg/600 mg (N=3) | Phase 1b Dose Escalation - 600 mg/800 mg (N=1) | Phase 1b Dose Escalation - 600 mg/1000 mg (N=1) | Phase 1b Dose Escalation - 600 mg (N=2) | Phase 1b Dose Escalation - 800 mg/1000 mg (N=5) | Phase 1b Dose Escalation - 800 mg (5 Days) (N=5) | Phase 1b Dose Escalation - 800 mg/600 mg (N=1) | Phase 1b Dose Escalation - 800 mg/800 mg (N=1) | Phase 1b Dose Escation - 800 mg (7 Days) (N=3) | Phase 2 - 800 mg/800 mg (N=27) | Phase 2 - 800 mg (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respirovirus test positive (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose Escalation - 600 mg/600 mg (N=3) | Phase 1b Dose Escalation - 600 mg/800 mg (N=1) | Phase 1b Dose Escalation - 600 mg/1000 mg (N=1) | Phase 1b Dose Escalation - 600 mg (N=2) | Phase 1b Dose Escalation - 800 mg/1000 mg (N=5) | Phase 1b Dose Escalation - 800 mg (5 Days) (N=5) | Phase 1b Dose Escalation - 800 mg/600 mg (N=1) | Phase 1b Dose Escalation - 800 mg/800 mg (N=1) | Phase 1b Dose Escation - 800 mg (7 Days) (N=3) | Phase 2 - 800 mg/800 mg (N=27) | Phase 2 - 800 mg (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT01790503/Prot_SAP_000.pdf